CLINICAL TRIAL: NCT02276573
Title: Study of Inflammatory Role of Epstein-Barr Virus (EBV) in Atrophic and Erosive Forms of Oral Lichen Planus
Acronym: LICHENVIR
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Centre Hospitalier Universitaire de Nice (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: 14-AOI-02
Record Dates: First submitted 2014-10-24; First posted 2014-10-28 (Estimated); Last update posted 2023-11-18 (Actual); Status verified 2023-11

CONDITIONS: Lichen Planus, Oral
MeSH Terms: conditions — Lichen Planus, Oral

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Oral lichen planus disease (Experimental): buccal cavity sample
  Interventions: Biological: buccal cavity sample

INTERVENTIONS:
Biological: buccal cavity sample

SUMMARY:
Oral lichen planus (OLP) is a chronic inflammatory and relapsing. The average prevalence is 1 to 4%. The clinics forms are many and symptoms are varied. The erosive form, painful and debilitating is characterized by erosive areas, ulcerated on an erythematous base with or without a keratinocyte lichenien network.

The literature data moving towards an autoimmune origin, but the pathophysiological mechanisms of OLP remain unknown.

This project represents the first part of a comprehensive project to examine the oral pathogenesis of different viruses (Herpes and papillomavirus HPV) and centered on Epstein-Barr Virus (EBV).

ELIGIBILITY:
Inclusion Criteria:

* Patient ≥ 18 years
* Clinical and/or histological diagnosis of erosive or atrophic OLP
* No signs of severe dysplasia at the sampling

Exclusion Criteria:

o immunosuppressive or anti-inflammatory therapies at the inclusion

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 13 (Actual)
Dates: Start 2015-03-30; Primary Completion 2016-03-10 (Actual); Study Completion 2016-03-10 (Actual)

PRIMARY OUTCOMES:
Measure of level of EBV nucleic acids | day 1

CONTACTS AND LOCATIONS:
Locations (1):
- Hôpital saint Roch, Nice, France

REFERENCES:
- [Derived] Raybaud H, Olivieri CV, Lupi-Pegurier L, Pagnotta S, Marsault R, Cardot-Leccia N, Doglio A. Epstein-Barr Virus-Infected Plasma Cells Infiltrate Erosive Oral Lichen Planus. J Dent Res. 2018 Dec;97(13):1494-1500. doi: 10.1177/0022034518788282. Epub 2018 Jul 13. PMID 30004820